CLINICAL TRIAL: NCT01744574
Title: Sex Differences & Progesterone: Association With Impulsivity and Smoking Cessation
Brief Title: Sex Differences, Hormones & Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2012NTLS074; P50DA033942-01 (NIH)
Record Dates: First submitted 2012-11-13; First posted 2012-12-06 (Estimated); Results first posted 2018-12-28 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Tobacco Cessation
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo - subjects will take 200 mg twice daily, orally (approximately 8am and 8pm) for twelve weeks starting seven days prior to the assigned quit date. They will also receive smoking cessation behavioral counseling.
  Interventions: Other: Placebo; Other: Smoking Cessation Behavioral Counseling
- Progesterone (Experimental): The progesterone will be given in the form of an active micronized natural progesterone (Prometrium). All subjects will take 200 mg twice daily, orally (approximately 8am and 8pm) for twelve weeks starting seven days prior to the assigned quit date. They will also receive smoking cessation behavioral counseling.
  Interventions: Drug: Progesterone; Other: Smoking Cessation Behavioral Counseling

INTERVENTIONS:
Other: Placebo — Placebo - subjects will take 200 mg twice daily orally (approximately 8am and 8pm) for twelve weeks starting seven days prior to the assigned quit date.
  Arms: Placebo
Drug: Progesterone — The progesterone will be given in the form of an active micronized natural progesterone (Prometrium). All subjects will take 200 mg twice daily orally (approximately 8am and 8pm) for twelve weeks starting seven days prior to the assigned quit date.
  Other Names: Prometrium
  Arms: Progesterone
Other: Smoking Cessation Behavioral Counseling — Subjects will receive weekly smoking cessation behavioral counseling.

SUMMARY:
Data suggest that progesterone may improve smoking cessation outcomes perhaps by reducing impulsive behavior. However, the clinical literature on this topic is lacking. Therefore, in Project I we are proposing a double-blind randomized controlled trial to assess the role of exogenous progesterone on impulsivity and smoking cessation in a sample of males and females who are motivated to quit smoking.

DETAILED DESCRIPTION:
Subjects will be stratified by sex and then randomly assigned to active progesterone (PRO) or placebo (PBO).

Telephone screening and visit invitation leads to the consent process and in-person screening including medical-psychiatric evaluation for inclusion/exclusion, then randomization and medication induction, stable medication with medication reduction and final evaluation for secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male 18 to 60 years old
* Female 18 to 50 years old
* Self-report regular smoking
* Motivated to quit smoking
* In stable physical/mental health
* Self report of regular menstrual cycles (female only)
* English fluency
* Understand the study procedures and able to provide informed consent
* Ability to participate fully in research elements for the duration of the trial.

Exclusion Criteria:

* Current or recent (< 3 months) breastfeeding (females only)
* Current or planned pregnancy within the next three months (females only)
* Conditions contraindicated to progesterone treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2012-12; Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon S. Allen, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Delaware Clinical Research Unit, University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo-Males; Placebo-Females: Placebo - subjects will take one placebo capsule twice daily, orally (approximately 8am and 8pm) for twelve weeks starting seven days prior to the assigned quit date. They will also receive smoking cessation behavioral counseling.
- Progesterone-Males; Progesterone-Females: Progesterone - The progesterone will be given in the form of an active micronized natural progesterone (Prometrium). Subjects will take 200 mg twice daily, orally (approximately 8am and 8pm) for twelve weeks starting seven days prior to the assigned quit date. They will also receive smoking cessation behavioral counseling.
Period: Overall Study
Arm/Group | Placebo-Males | Progesterone-Males | Placebo-Females | Progesterone-Females
Started | 57 | 56 | 52 | 51
Completed | 33 | 31 | 32 | 40
Not Completed | 24 | 25 | 20 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo-Males | Progesterone-Males | Placebo-Females | Progesterone-Females | Total
Number analyzed (Participants) | 57 | 56 | 52 | 51 | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (11.8) | 37.9 (10.6) | 36.0 (7.8) | 37.6 (7.4) | 37.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 52 | 51 | 103
  Male | 57 | 56 | 0 | 0 | 113
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race (non-white) | 25 | 22 | 21 | 20 | 88
  Race (white) | 32 | 34 | 31 | 31 | 128

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 7-day Point Prevalence Abstinence From Smoking at Week 4
Description: 7-day point prevalence abstinence from smoking defined as having no slips (i.e., a puff or more from a lit cigarette) in the seven days prior to week 4
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Males | Progesterone-Males | Placebo-Females | Progesterone-Females
Number analyzed (Participants) | 57 | 56 | 52 | 51
Participants | 12 | 13 | 9 | 18

2. Secondary Outcome: Number of Participants With 7-day Point Prevalence Abstinence From Smoking at Weeks 8 and 12
Description: 7-day point prevalence abstinence from smoking defined as having no slips (i.e., a puff or more from a lit cigarette) in the seven days prior to weeks 8 and 12
Time Frame: Weeks 8 and 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Males | Progesterone-Males | Placebo-Females | Progesterone-Females
Number analyzed (Participants) | 57 | 56 | 52 | 51
Participants
  Week 8 | 10 | 10 | 10 | 16
  Week 12 | 12 | 7 | 12 | 20

3. Secondary Outcome: Number of Participants With Prolonged Abstinence From Smoking at Weeks 4, 8 and 12
Description: Prolonged abstinence defined as having less than seven consecutive slips without a 24-hour period between any two slips prior to weeks 4, 8 and 12
Time Frame: Weeks 4, 8 and 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Males | Progesterone-Males | Placebo-Females | Progesterone-Females
Number analyzed (Participants) | 57 | 56 | 52 | 51
Participants
  Week 4 | 15 | 11 | 10 | 18
  Week 8 | 9 | 7 | 8 | 15
  Week 12 | 7 | 6 | 7 | 13

4. Secondary Outcome: Number of Participants With Continuous Abstinence From Smoking at Week 12
Description: continuous abstinence defined as having no slips at all prior to week 12
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Males | Progesterone-Males | Placebo-Females | Progesterone-Females
Number analyzed (Participants) | 57 | 56 | 52 | 51
Participants | 4 | 4 | 2 | 8

5. Secondary Outcome: Number of Participants With Cotinine <50 ng/mL at Weeks 4, 8 and 12
Description: urine cotinine <50 ng/mL at weeks 4, 8 and 12
Time Frame: Weeks 4, 8 and 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Males | Progesterone-Males | Placebo-Females | Progesterone-Females
Number analyzed (Participants) | 57 | 56 | 52 | 51
Participants
  Week 4 | 9 | 11 | 8 | 10
  Week 8 | 7 | 8 | 8 | 10
  Week 12 | 6 | 9 | 9 | 10

6. Secondary Outcome: Number of Participants With Breath Carbon Monoxide ≤5 Ppm at Weeks 4, 8 and 12
Description: breath carbon monoxide ≤5 ppm at weeks 4, 8 and 12
Time Frame: Weeks 4, 8 and 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Males | Progesterone-Males | Placebo-Females | Progesterone-Females
Number analyzed (Participants) | 57 | 56 | 52 | 51
Participants
  Week 4 | 17 | 20 | 18 | 22
  Week 8 | 14 | 13 | 16 | 17
  Week 12 | 9 | 14 | 20 | 19

7. Secondary Outcome: Average Number of Days to Relapse
Description: Days to relapse defined as the number of days from quit date to the first day with a slip
Time Frame: Days 1 through 84
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo-Males | Progesterone-Males | Placebo-Females | Progesterone-Females
Number analyzed (Participants) | 57 | 56 | 52 | 51
days | 13.3 (23.8) | 13.4 (25.9) | 14.3 (26.8) | 20.5 (29.6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected between enrollment and study completion (or study dropout) which ever came first; an average of 16 weeks .
Arm/Group | Placebo-Males | Progesterone-Males | Placebo-Females | Progesterone-Females
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/56 | 0/52 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/57 | 1/56 | 0/52 | 0/51
Other Adverse Events (participants affected / at risk) | 0/57 | 0/56 | 0/52 | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-Males (N=57) | Progesterone-Males (N=56) | Placebo-Females (N=52) | Progesterone-Females (N=51)
Stroke (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Generalizability is limited as our sample included only premenopausal women. The sample size was too small to directly compare sex differences between men and women. Participants were only followed for 12 weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT01744574/Prot_SAP_000.pdf